CLINICAL TRIAL: NCT04911530
Title: Perioperative Database of Chinese Elderly Patients
Acronym: PDCEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); Peking University First Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Xiangya Hospital of Central South University (Other); Beijing Anzhen Hospital (Other); Central South University (Other); Peking University People's Hospital (Other); Zhejiang University (Other); Fudan University (Other); Sun Yat-sen University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); China-Japan Friendship Hospital (Other); The Affiliated Hospital Of Guizhou Medical University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Taihe Hospital (Other); Zhejiang Provincial People's Hospital (Other); Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director, Department of Anesthesiology (Cheif expert of National key research and development program of China 2018YFC2001900), Chinese PLA General Hospital
Other Study IDs: PLAGH-AOC-001
Record Dates: First submitted 2021-03-28; First posted 2021-06-03 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Perioperative Complications; Perioperative/Postoperative Complications; Perioperative Adverse Events
Keywords: central nervous system complications; heart injury; acute kidney injury; lung injury; infection; pain
MeSH Terms: conditions — Postoperative Complications; Heart Injuries; Acute Kidney Injury; Lung Injury; Infections; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- elderly patients (aged ≥ 65 years): elderly patients undergo surgeries
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The investigators aim to establish a prospective database of perioperative elderly patients from multiple regions and centers. Collected data involves postoperative complications of the central nervous system, cardiovascular system, kidney, respiratory system, infection, pain, and other perioperative complications. Based on the database, the investigators intend to explore:

* The incidence and risk factors of perioperative morbidity and mortality in elderly patients;
* Perioperative risk assessment methods and early warning models for elderly patients;
* Practical, safe, and effective risk prevention and control system through subsequent studies.

DETAILED DESCRIPTION:
As the population aging is speeding up, senile diseases have become a significant and severe public health problem, influencing national health. More than 20 million elderly patients undergo surgery each year in China, accounting for a quarter of the population who undergo surgery. Advanced age and comorbid diseases render the elderly at increased risk of postoperative morbidity and mortality. The incidence of postoperative complications is twice that of non-elderly patients, and mortality rates are five times higher than non-elderly patients. Thus, it is a significant challenge to safely and stably ensure the elderly are in an optimal perioperative period.

For the good of optimizing perioperative management, it is urgent to build a large-sample, multi-center database. Based on this database, the investigators can explore new risk assessment methods and establish a perioperative risk prediction model and early warning system suitable for elderly patients. It will help improve this group of patients' short- and long-term outcomes and thus reduce the economic burden of national health and medical resources.

In this context, establishing a clinical database including data for all perioperative elderly patients is of high interest. This database will allow the investigators to carry out clinical research on:

* Clinical, biological, and genetic factors predictive of perioperative complications and deaths;
* Systematic and individualized evaluation tools for elderly patients;
* Prognostic factors for improving short- and long-term outcomes. This is particularly significant for rare clinical evidence of perioperative elderly patients for which the current knowledge is scarce.

The database will also allow the investigators to develop or participate in multi-center trials, national or international, and facilitate the formation of perioperative data collection standards.

ELIGIBILITY:
Inclusion Criteria:

* Geriatric surgical patients ≥65 years old, undergoing elective surgery with a planned overnight hospital stay following surgery.

Exclusion Criteria:

* Patients fully refused to participate in the study;
* Patients with severe dementia, language disorder, severe hearing or visual impairment, coma, and end-stage status were excluded;
* Patients whose surgeries were canceled;
* Patients accepted cardiac surgeries were excluded from the heart injury section;
* Patients accepted cardiac, neurosurgeries or were excluded from postoperative central nervous system and pain observation section;
* Patients refused to participate in neurocognitive, anxiety, depression, or pain questionnaire were excluded from relative assessment and measurement.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Hospital-based, elderly patients, perioperative/postoperative outcome/complications study
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | Up to 30 days
  Clinical data of postoperative complications in the medical record and follow-up update. Postoperative complications, including central nervous system injury, heart injury, acute kidney injury, lung injury, infection, and pain.
Postoperative Survival | Up to 30 days
  Clinical data of survival in the medical record and follow-up update.

OTHER OUTCOMES:
Postoperative Survival | 1 year after surgeries
  Clinical data of survival in the medical record and follow-up update.
Postoperative complications | 1 year after surgeries
  Clinical data of postoperative complications in the medical record and follow-up update. Postoperative complications, including central nervous system injury, heart injury, acute kidney injury, lung injury, infection, and pain.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Mi, PhD, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided